CLINICAL TRIAL: NCT06935968
Title: Effect of Levonorgestrel Intrautrine System on Hemoglobin Level and Iron Profile on Women Requiring Contraception
Brief Title: Effect of Levonorgestrel Intrauterine System on Hemoglobin Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Melad Matta, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Mirena
Record Dates: First submitted 2025-04-07; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hemoglobin; Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel intrauterine system insertion (Other)
  Interventions: Device: Levonorgestrel intrautrine system

INTERVENTIONS:
Device: Levonorgestrel intrautrine system — Insertion of levonorgestrel intrautrine system and take a blood sample from the women to analyse it
  Other Names: Take a blood sample

SUMMARY:
To study the effect of LNG-IUS on improving iron status in reproductive-aged women presenting for contraception.

DETAILED DESCRIPTION:
Women come to family planning clinic to insert levonorgestrel intrautrine system and take a blood sample from her to analyse hemoglobin level

ELIGIBILITY:
Inclusion Criteria:

1. The study will include married women attending the outpatient clinics of the forementioned health facilities for contraception counseling
2. Age between 18 and 45 years
3. Women who choose LNG_IUS for contraception
4. Any parity including nulliparous

Exclusion Criteria:

* 1.Women with any inherited hemoglobinopathy (thalassemia, sickle cell anemia) or acquired hemolytic anemia 2.Women with sever iron deficiency anemia requiring immediate treatment 3.Women with any contraindication to Mirena insertion (pelvic inflammatory disease, cervical or vaginal infection, cervical cancer) 4. Any uterine abnormality making LNG_IUS insertion difficult (septate uterus or fibroid distorting the cavity) 5. Women within 6 months of delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change of blood haemoglobin level from time of insertion to 6 months after insertion | 6 months
  To know the effect of LNG-IUDs on hemoglobin level after insertion

SECONDARY OUTCOMES:
Change of serum ferritin level from time of insertion to 6 months after insertionPrevalence of iron deficiency and iron deficiency anemia in women requiring contraception in our community | 6 months
  To know the effect of LNG-IUDs in serum ferritin